CLINICAL TRIAL: NCT01341327
Title: A GLOBAL, MULTICENTER, PROSPECTIVE, REAL WORLD OBSERVATIONAL STUDY FOR LEFT MAIN DISEASE TREATMENT
Brief Title: Observational Study for Left Main Disease Treatment
Acronym: IRIS-MAIN
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2010-08
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
Keywords: Left Main
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Left Main disease: Consecutive patients with unprotected LMCA diseases at participating centers will be evaluated for the entry into the study.

SUMMARY:
The purpose of this study is to observe clinical courses for long-term in patients with unprotected LMCA disease and to evaluate comparative results of medical treatment, coronary stenting with drug-eluting stents, and CABG for the treatment of an unprotected LMCA stenosis in the "real world" daily practice.

DETAILED DESCRIPTION:
This study is a multicenter, large clinical registry to evaluate comparative outcomes of medical therapy, PCI with DES, or CABG for patients with unprotected LMCA stenosis in the Asia-Pacific, as recorded in the MAIN-IRIS Registry. Data will be prospectively collected on approximately 5000 subjects who diagnosed LM disease (>50% by visual estimation) at approximately 65 centers in Korea and Asia-Pacific region. Brief study design is as depicted in the following figure

ELIGIBILITY:
Inclusion Criteria:

* Significant unprotected left main stenosis (>50% by visual estimation)

  * The LMCA is considered unprotected if there are no patent coronary artery bypass grafts to the left anterior descending artery or the left circumflex artery.
* No limitation of clinical or lesion characteristics
* Age >18 years
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Protected left main stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with unprotected LMCA diseases at participating centers will be evaluated for the entry into the study.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2007-07 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Composite event rate of death, myocardial infarction, Target Vessel Revascularization or cerebrovascular event | 2-year
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
Death | 10-year
Cardiac death | 10-year
Myocardial infarction | 10-year
Cerebrovascular event | 10-year
Target vessel revascularization | 10-year
Target lesion revascularization | 10-year
Stent thrombosis | 10-year
  According to Academic Research Consortium (ARC) criteria
Binary restenosis and late luminal loss in both in-stent and in-segment | 9-month
  Angiographic follow-up in the PCI group (as form of PCI substudy)
Rehospitalization | 10-year

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — CVRF
Locations (42):
- Zhongshan Hospital, Shanghai, China
- Sarawak General Hospital, Kuching, Malaysia
- South Korea (38):
  - Hallym University medical center, Anyang
  - Soonchunhyang University Hospital, Buchen, Bucheon-si
  - The Catholic University of Korea, Bucheon ST.Mary's Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Soonchunhyang University Hospital, Cheonan, Cheonan
  - St.Mary's Catholic Medical Center, Cheongju-si
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST.Mary's Hospital, Daejeon
  - Gangneung Asan Medical Center, Gangneung
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - St.Mary's Catholic Medical Center, Inchon
  - Chonbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Kwangju Christian hospital, Kwangju
  - Pusan Natioanal University Hospital, Pusan
  - Bundang CHA Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Dongguk University Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangbuk samsung hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Anam hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - St.Mary's Catholic Medical Center, Seoul
  - The Catholic University of Korea, ST. Paul's Hospital, Seoul
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul
  - Yonsei University Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Christian Hospital, Wŏnju
- Shin Kong Hospital, Taipei, Taiwan
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial

REFERENCES:
- [Derived] Kim TO, Kang DY, Ahn JM, Kim MJ, Lee PH, Kim H, Choi Y, Lee J, Lee JM, Jo HH, Park YS, Lim SM, Park SJ, Park DW. Impact of Target Lesion Revascularization on Long-Term Mortality After Percutaneous Coronary Intervention for Left Main Disease. JACC Cardiovasc Interv. 2024 Jan 8;17(1):32-42. doi: 10.1016/j.jcin.2023.10.068. PMID 38199751
- [Derived] Cho S, Kang DY, Kim JS, Park DW, Kim IS, Kang TS, Ahn JM, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Lee SJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Jang Y, Hong MK, Park SJ. Dual antiplatelet therapy after percutaneous coronary intervention for left main coronary artery disease. Rev Esp Cardiol (Engl Ed). 2023 Apr;76(4):245-252. doi: 10.1016/j.rec.2022.07.007. Epub 2022 Jul 27. English, Spanish. PMID 35907438
- [Derived] Park S, Ahn JM, Park H, Kang DY, Lee PH, Kim TO, Lee J, Kim JH, Yang Y, Jeong YJ, Hyun J, Kim AR, Kim T, Oh HJ, Lee YJ, Lee JH, Jang M, Park DW, Park SJ; IRIS-MAIN Registry Investigators. Comparison of Long-Term Outcomes Following Coronary Revascularization in Men-vs-Women with Unprotected Left Main Disease. Am J Cardiol. 2021 Aug 15;153:9-19. doi: 10.1016/j.amjcard.2021.05.016. Epub 2021 Jul 4. PMID 34233836
- [Derived] Park S, Ahn JM, Kim TO, Park H, Kang DY, Lee PH, Jeong YJ, Hyun J, Lee J, Kim JH, Yang Y, Choe K, Park SJ, Park DW; IRIS-MAIN Registry Investigators. Revascularization in Patients With Left Main Coronary Artery Disease and Left Ventricular Dysfunction. J Am Coll Cardiol. 2020 Sep 22;76(12):1395-1406. doi: 10.1016/j.jacc.2020.07.047. PMID 32943156
- [Derived] Kang SH, Ahn JM, Lee CH, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park DW, Park SJ. Differential Event Rates and Independent Predictors of Long-Term Major Cardiovascular Events and Death in 5795 Patients With Unprotected Left Main Coronary Artery Disease Treated With Stents, Bypass Surgery, or Medication: Insights From a Large International Multicenter Registry. Circ Cardiovasc Interv. 2017 Jul;10(7):e004988. doi: 10.1161/CIRCINTERVENTIONS.116.004988. PMID 28701487